CLINICAL TRIAL: NCT03194685
Title: A First-in-Human Phase 1 Study to Assess the Safety, Tolerability, Efficacy, and Pharmacokinetics of FF-10101-01 in Subjects With Relapsed or Refractory Acute Myeloid Leukemia
Brief Title: Study of FF-10101-01 in Patients With Relapsed or Refractory Acute Myeloid Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fujifilm Pharmaceuticals U.S.A., Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: FF-10101-US101
Record Dates: First submitted 2017-05-04; First posted 2017-06-21 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: AML, Adult
Keywords: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Cohort 1: 10 mg (Experimental): Orally once a day (QD) on Days 1-28 of a 28-day cycle. Drug: FF-10101-01
  Interventions: Drug: FF-10101-01
- Cohort 2: 20 mg (Experimental): Orally once a day (QD) on Days 1-28 of a 28-day cycle. Drug: FF-10101-01
  Interventions: Drug: FF-10101-01
- Cohort 3: 35 mg (Experimental): Orally once a day (QD) on Days 1-28 of a 28-day cycle. Drug: FF-10101-01
  Interventions: Drug: FF-10101-01
- Cohort 4: 50 mg (Experimental): Orally once a day (QD) on Days 1-28 of a 28-day cycle. Drug: FF-10101-01
  Interventions: Drug: FF-10101-01
- Cohort 5: 75 mg (Experimental): Orally once a day (QD) on Days 1-28 of a 28-day cycle. Drug: FF-10101-01
  Interventions: Drug: FF-10101-01
- Cohort 6: 100 mg (Experimental): Orally once a day (QD) on Days 1-28 of a 28-day cycle. Drug: FF-10101-01
  Interventions: Drug: FF-10101-01
- Cohort 7: 150 mg (Experimental): Orally once a day (QD) on Days 1-28 of a 28-day cycle. Drug: FF-10101-01
  Interventions: Drug: FF-10101-01
- Cohort 8: 225 mg (Experimental): Orally once a day (QD) on Days 1-28 of a 28-day cycle. Drug: FF-10101-01
  Interventions: Drug: FF-10101-01

INTERVENTIONS:
Drug: FF-10101-01 — FF-10101-01 will be administered orally once a day on Days 1-28 of a 28-day cycle. In Phase 1, the dose escalation will proceed until MTD is reached.
  Other Names: FF-10101 succinate

SUMMARY:
A Phase 1 dose escalation and dose ranging study of FF-10101-01 in subjects with relapsed or refractory acute myeloid leukemia to determine the safety, tolerability, PK and preliminary efficacy. A total of 9 cohorts will be enrolled in Phase 1 to establish the Maximum Tolerated Dose (MTD).

DETAILED DESCRIPTION:
Subjects will receive FF-10101-01 orally once a day repeated every 28 days =1 cycle Frequent blood draws will be collected to measure pharmacodynamic parameters and pharmacodynamic activity.

Disease assessments, including bone marrow aspirates, will be performed at the beginning of cycles 1-3, and every 3 months thereafter. Subjects who demonstrate objective response or stable disease will be allowed to continue therapy with FF-10101-01 until , observation of unacceptable adverse events, or until the subject is no longer deriving benefit based on the opinion of the investigator.

ELIGIBILITY:
Subjects who are able and willing to give written informed consent

* Documented primary or secondary AML, as defined by the WHO criteria (2008), by histopathology refractory to previous induction chemotherapy and/or relapsed after achieving remission with a prior chemotherapy and who are not candidates for other available therapy likely to confer clinical benefit.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2
* In the absence of rapidly progressing disease, the interval from prior treatment to time of FF-10101-01 administration should be at least 14 days for cytotoxic agents other than hydroxyurea, at least 5 half-lives for non-cytotoxic agents, and 14 days for monoclonal antibody therapies. Hydroxyurea may be continued for a maximum of 14 days from the start of FF-10101-01 dosing, through Cycle 1 Day 14, with a maximal dose of 5 grams/day
* Persistent chronic clinically significant toxicities from prior chemotherapy or surgery must be ≤Grade 2
* If subject has had a hematopoietic stem cell transplant, subject must be ≥60 days post-transplant with no clinically significant GVHD requiring systemic therapy
* Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) ≤3 times the upper limit of normal and total bilirubin of ≤1.5x the upper limit of normal. If total bilirubin is equal to or exceeds 1.5x the upper limit of normal, the subject can still be included if direct bilirubin is ≤1.5x the upper limit of normal
* Calculated creatinine clearance of ≥60 mL/min
* Female subjects of childbearing potential and sexually mature male subjects must agree to use a medically accepted method of contraception other than an oral contraceptive for the duration of the study.

Exclusion Criteria:

* Subjects diagnosed with acute promyelocytic leukemia
* Subjects with Bcr-Abl positive leukemia (chronic myelogenous leukemia in blast crisis)
* Subjects with clinically active CNS leukemia
* Subjects with major surgery within 28 days prior to the first administration of FF-10101-01
* Subjects with radiation therapy within 28 days prior to the first administration of FF-10101-01
* Subjects with active malignant disease requiring therapy other than AML or myelodysplastic syndrome with transformation into AML
* Subjects with an active uncontrolled infection
* Subjects with a medical condition, serious intercurrent illness, or other circumstance that, in the Investigator's judgment, could jeopardize the subject's safety as a study subject, or that could interfere with the study objectives
* Subjects known to have human immunodeficiency virus infection, or who have active hepatitis B or C infection as determined by serological testing
* Subjects with congestive heart failure, New York Heart Association (NYHA) Class 3 or 4, or subjects with a past history of congestive heart failure NYHA Class 3 or 4 and in whom echocardiogram or multiple gate acquisition (MUGA) scan performed within 3 months prior to screening or at screening showed a LVEF <40%
* Female subjects who are pregnant or breast feeding
* Subjects on 3-hydroxy-3-methylglutaryl-coenzyme A reductase inhibitors (statins) or other drugs known to have muscle toxicity
* Subjects taking strong inhibitors of CYP3A4 will be excluded from the study unless therapeutic substitution is possible
* Subjects taking strong inducers of CYP3A4 will be excluded from the study unless therapeutic substitution is possible
* Use of systemic immunosuppressive agents within 14 days prior to first dose of FF-10101
* Subjects taking drugs known to cause Torsades de Pointes will be excluded from the study unless therapeutic substitution is possible
* Subjects known to have long QT syndrome
* Subjects with mean QTcF values following 3 ECGs conducted 5 minutes apart of >470 msec

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2017-05-05 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Phase 1: Frequency of adverse events | 12 months
  Safety Assessments include frequency of adverse events (AEs) in percentage (%)

SECONDARY OUTCOMES:
Phase 1: Evaluate the Pharmacokinetic profile of FF-10101-01 and its Metabolite - Maximum observed concentration (Cmax) | Cycle 1, Day 1 through Cycle 2, Day 1
  Maximum observed concentration (Cmax)
Phase 1: Evaluate the Pharmacokinetic profile of FF-10101-01 and its Metabolite - Time to maximum concentration (tmax) | Cycle 1, Day 1 through Cycle 2, Day 1
  Time to maximum concentration (tmax)
Phase 1: Evaluate the Pharmacokinetic profile of FF-10101-01 and its Metabolite - Area under the plasma concentration-time curve in the sampled matrix during a 24-hour dosing interval (AUC(τ)) | Cycle 1, Day 1 through Cycle 2, Day 1
  Area under the plasma concentration-time curve in the sampled matrix during a 24-hour dosing interval (AUC(τ))
Phase 1: Evaluate the Pharmacokinetic profile of FF-10101-01 and its Metabolite -Plasma concentration-time curve (AUC(0-last)) | Cycle 1, Day 1 through Cycle 2, Day 1
  Area under the plasma concentration-time curve in the sampled matrix from time zero to the last quantifiable concentration, if concentrations are not quantifiable over the entire 24-hour dosing interval (AUC(0-last))
Phase 1: Evaluate the Pharmacokinetic profile of FF-10101-01 and its Metabolite - Dose normalized AUC(τ) (AUC(τ)/dose) | Cycle 1, Day 1 through Cycle 2, Day 1
  Dose normalized AUC(τ) (AUC(τ)/dose)
Phase 1: Evaluate the Pharmacokinetic profile of FF-10101-01 and its Metabolite - Dose normalized Cmax (Cmax/dose) | Cycle 1, Day 1 through Cycle 2, Day 1
  Dose normalized Cmax (Cmax/dose)
Phase 1: Evaluate the Pharmacokinetic profile of FF-10101-01 and its Metabolite - Accumulation ratio for AUC | Cycle 1, Day 1 through Cycle 2, Day 1
  Accumulation ratio for AUC [RaccAUC ie, ratio of Day 29/Day 1 of the PK parameter]
Phase 1: Evaluate the Pharmacokinetic profile of FF-10101-01 and its Metabolite - Accumulation ratio for Cmax | Cycle 1, Day 1 through Cycle 2, Day 1
  Accumulation ratio for Cmax [RaccCmax ie, ratio of Day 29/Day 1 of the PK parameter]
Phase 1: Evaluate the Pharmacokinetic profile of FF-10101-01 and its Metabolite - Oral clearance (CL/F) for FF-10101 | Cycle 1, Day 1 through Cycle 2, Day 1
  Oral clearance (CL/F) for FF-10101
Phase 1: Evaluate the Pharmacokinetic profile of FF-10101-01 and its Metabolite - Average concentrations (Cavg) | Cycle 1, Day 1 through Cycle 2, Day 1
  Average concentrations (Cavg)
Phase 1: Evaluate the Pharmacokinetic profile of FF-10101-01 and its Metabolite - Minimum observed concentration (Cmin) | Cycle 1, Day 1 through Cycle 2, Day 1
  Minimum observed concentration (Cmin)
Phase 1: Evaluate the Pharmacokinetic profile of FF-10101-01 and its Metabolite - Fluctuation index | Cycle 1, Day 1 through Cycle 2, Day 1
  Fluctuation index
Phase 1: Evaluate the Pharmacokinetic profile of FF-10101-01 and its Metabolite - Metabolite (FF-10101M1) to parent (FF-10101) exposure ratios for Cmax | Cycle 1, Day 1 through Cycle 2, Day 1
  Metabolite (FF-10101M1) to parent (FF-10101) exposure ratios for Cmax
Phase 1: Evaluate the Pharmacokinetic profile of FF-10101-01 and its Metabolite - Metabolite (FF-10101M1) to parent (FF-10101) exposure ratios for AUC(τ) | Cycle 1, Day 1 through Cycle 2, Day 1
  Metabolite (FF-10101M1) to parent (FF-10101) exposure ratios for AUC(τ)
Phase 1: Frequency of Serious Adverse Events | 12 Months
  Safety Assessments include frequency of Serious adverse events (SAEs)
Phase 1: Frequency of Dose Limiting Toxicities | 12 Months
  Safety Assessments include frequency of dose-limiting toxicities (DLTs), dose reductions, delays, or withdrawals due to toxicity.
Phase 1: Frequency of adverse events including assessment of Hematology laboratory parameters | 12 Months
  Safety assessments also include assessment of clinical laboratory parameters Hematology
Phase 1: Frequency of adverse events including assessment of serum chemistry laboratory parameters | 12 Months
  Safety assessments also include assessment of clinical laboratory parameters serum chemistry
Phase 1: Frequency of adverse events including assessment of urinalysis laboratory parameters | 12 Months
  Safety assessments also include assessment of clinical laboratory parameters urinalysis
Phase 1: Frequency of Adverse events including assessment of vital signs | 12 Months
  Safety assessments also include assessment of Vital signs (Heart Rate and BP)
Phase 1: Frequency of Adverse events including assessment of vital signs - Heart Rate | 12 Months
  Safety assessments also include assessment of Vital signs Heart Rate
Phase 1: Frequency of Adverse events including assessment of vital signs - Blood Pressure | 12 Months
  Safety assessments also include assessment of Vital signs BP)
Phase 1: Frequency of Adverse events including assessment of 12 lead ECG. | 12 Months
  Safety assessments also include assessment of 12 lead ECG.
Phase 1: Composite complete remission rate (CRc) including CR | 12 Months
  Composite complete remission rate (CRc) which includes CR
Phase 1: Composite complete remission rate (CRc) including CR with incomplete platelet recovery (CRp) | 12 Months
  Composite complete remission rate (CRc) which includes CR with incomplete platelet recovery (CRp)
Phase 1: Composite complete remission rate (CRc) including CR with incomplete neutrophil recovery with or without platelet recovery (CRi)) | 12 Months
  Composite complete remission rate (CRc) which includes CR with incomplete neutrophil recovery with or without platelet recovery (CRi))

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - University of California Los Angeles, David Geffen School of Medicine, Los Angeles, California
  - University Of California, San Francisco School of Medicine, San Francisco, California
  - Northwestern University, Chicago, Illinois
  - Johns Hopkins Hospital - Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Levis M, Perl A, Schiller G, Fathi AT, Roboz G, Wang ES, Altman J, Rajkhowa T, Ando M, Suzuki T, Subach RA, Maier G, Madden T, Johansen M, Cheung K, Kurman M, Smith C. A phase 1 study of the irreversible FLT3 inhibitor FF-10101 in relapsed or refractory acute myeloid leukemia. Blood Adv. 2024 May 28;8(10):2527-2535. doi: 10.1182/bloodadvances.2023010619. PMID 38502195